CLINICAL TRIAL: NCT00874757
Title: Effect of Rosuvastatin Response in Healthy Subjects: Potential Mechanisms of
Brief Title: Effect of Rosuvastatin Response in Healthy Subjects: Potential Mechanisms of Anti-inflammatory Effects
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0088-09-FB
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Statins, anti-inflammatory; Healthy subjects study
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rosuvastatin: Healthy subjects received rosuvastatin 20 mg orally for 3 weeks. Inflammatory markers measured pre and post rosuvastatin treatment.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Healthy subjects received rosuvastatin 20 mg orally for 3 weeks. Inflammatory markers measured pre- and post- rosuvastatin treatment.
  Other Names: Crestor

SUMMARY:
The purpose of this study is to see whether Statin drugs will act as anti-inflammatories. The investigators will study this potential anti-inflammatory activity in healthy subjects.

DETAILED DESCRIPTION:
After providing consent healthy subjects (N=20) completed a health and drug inventory questionnaire and had blood samples drawn to measure baseline electrolytes, kidney function, liver function, and creatine kinase to determine study eligibility. Blood samples were also collected to analyze baseline inflammatory markers (tlr-4 monocyte expression and cytokine production). Patients received 20 mg daily of rosuvastatin for 3 weeks followed by blood collection, and the measurement of inflammatory markers repeated. Whole blood samples were analyzed by flow-cytometry to determine percent expression of tlr-4 on monocytes which was the primary inflammatory marker for the study. Secondary inflammatory markers tumor necrosis factor (TNF), interleukin-6 (IL-6), and interleukin-8 (IL-8) were measured after blood was incubated ex-vivo with lipopolysaccharide (LPS) for 3 hours. LPS induction experiments were performed on blood from pre and post rosuvastatin treatment. Finally, blood lipid profiles (cholesterol, low density lipoprotein (LDL), very low-density lipoprotein (VLDL), and high density lipo protein (HDL), were assessed both pre and post rosuvastatin treatment. End of study (after 3 weeks of rosuvastatin treatment) electrolytes, kidney function, liver function, and creatine kinase (CK) were measured to determine any changes as a result of rosuvastatin treatment. In addition to pre and post safety assessment a phone call was made to evaluate rosuvastatin side effects at the midpoint of the three-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male non-asian subjects

Exclusion Criteria:

* Patients with increased liver function tests, elevated serum creatine, patients on anti-inflammatory or immunomodulating drugs

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R McGuire, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Pharmacy, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wickelgren I. Immunology. Targeting the tolls. Science. 2006 Apr 14;312(5771):184-7. doi: 10.1126/science.312.5771.184. No abstract available. PMID 16614188
- [Background] Falagas ME, Makris GC, Matthaiou DK, Rafailidis PI. Statins for infection and sepsis: a systematic review of the clinical evidence. J Antimicrob Chemother. 2008 Apr;61(4):774-85. doi: 10.1093/jac/dkn019. Epub 2008 Feb 7. PMID 18263570
- [Background] Niessner A, Steiner S, Speidl WS, Pleiner J, Seidinger D, Maurer G, Goronzy JJ, Weyand CM, Kopp CW, Huber K, Wolzt M, Wojta J. Simvastatin suppresses endotoxin-induced upregulation of toll-like receptors 4 and 2 in vivo. Atherosclerosis. 2006 Dec;189(2):408-13. doi: 10.1016/j.atherosclerosis.2005.12.022. Epub 2006 Jan 26. PMID 16443229
- [Background] Novack V, Eisinger M, Frenkel A, Terblanche M, Adhikari NK, Douvdevani A, Amichay D, Almog Y. The effects of statin therapy on inflammatory cytokines in patients with bacterial infections: a randomized double-blind placebo controlled clinical trial. Intensive Care Med. 2009 Jul;35(7):1255-60. doi: 10.1007/s00134-009-1429-0. Epub 2009 Feb 11. PMID 19205663
- [Background] Wang CY, Liu PY, Liao JK. Pleiotropic effects of statin therapy: molecular mechanisms and clinical results. Trends Mol Med. 2008 Jan;14(1):37-44. doi: 10.1016/j.molmed.2007.11.004. PMID 18068482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 subjects were consented between 11/15/2010 and on 8/4/2011.
Groups:
- Rosuvastatin: 20 subjects were consented to receive rosuvastatin 20 mg tablets orally every day for three weeks. 16 of the 20 received study drug with four being excluded due to baseline laboratory abnormalities.
Period: Overall Study
Arm/Group | Rosuvastatin
Started | 20 (Institutional review board (IRB) approved consents on 11-11-2010 with first subject consented on 11-15-2010)
Completed | 16 (While 20 subjects were consented 3 subjects were excluded from receiving rosuvastatin based on elevated liver function tests and 1 subject based on elevated creatine kinase.)
Not Completed | 4
Not completed — Baseline laboratories outside of normal limits (screen fails). | 4

BASELINE CHARACTERISTICS:
Population: The 16 patients that met inclusion/exclusion criteria were Caucasian.
Groups:
- Rosuvastatin: Single arm non-therapeutic study where all subjects who ruled in for study participation (based on baseline laboratories and clinical assessment) received rosuvastatin 20 mg tablets for three weeks. Inflammatory markers Toll-like Receptor 4, tumor necrosis factor, Interleukin 6, Interleukin 8 (tlr-4, TNF, IL-6, IL-8) were measured at baseline prior to rosuvastatin administration and after treatment to compare the effect of rosuvastatin on inflammatory markers. The primary outcome was the %tlr positive monocytes.
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 27 [22 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Toll-like Receptor 4 Expression Pre- and Post-Treatment
Description: Toll-like Receptor 4 (TLR-4) expression on monocytes in whole blood pre- and post- 3 weeks of rosuvastatin treatment.
Time Frame: Before and after three weeks of treatment with rosuvastatin
Population: A total of 16 healthy subjects who met inclusion/exclusion criteria
Measure: Mean (Standard Deviation); unit: % tlr expression (monocytes)
Groups:
- Pre-treatment Tlr-4 Expression: Whole blood collected analyzed by flow cytometry prior to the start of rosuvastatin
- Post-treatment Trl-4 Monocyte Expression: Flow cytometry performed on blood after 3 weeks of treatment with rosuvastatin
Arm/Group | Pre-treatment Tlr-4 Expression | Post-treatment Trl-4 Monocyte Expression
Number analyzed (Participants) | 16 | 16
% tlr expression (monocytes) | 12.37 (9.8) | 6.36 (4.8)

2. Secondary Outcome: Tumor Necrosis Factor (TNF)
Description: Inflammatory cytokine generated after treatment of whole blood collected before and after rosuvastatin treatment
Time Frame: Pre and post 3 weeks of rosuvastatin treatment
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Baseline (Pre-Rosuvastatin Treatment): 16 subjects had blood collected before treatment with rosuvastatin and blood was treated with LPS ex-vivo and TNF concentrations measured.
- Post Rosuvastatin Treatment: Blood samples collected were treated with Lipopolysaccharides (LPS) and tumor necrosis factor (TNF) measured
Arm/Group | Baseline (Pre-Rosuvastatin Treatment) | Post Rosuvastatin Treatment
Number analyzed (Participants) | 16 | 16
pg/ml | 145 (52) | 92 (25)

3. Secondary Outcome: Interleukin-6
Description: Interleukin-6 inflammatory cytokine which will be released after LPS treatment of blood
Time Frame: Before (baseline) and after 3 weeks of rosuvastatin treatment
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Interleukin-6 Baseline (Before Rosuvastatin Treatment): Interleukin-6 concentrations after blood treated with LPS (baseline)
- Interleukin-6 Post-treatment: Interleukin-6 concentrations after blood treated with LPS after 3 weeks of rosuvastatin
Arm/Group | Interleukin-6 Baseline (Before Rosuvastatin Treatment) | Interleukin-6 Post-treatment
Number analyzed (Participants) | 16 | 16
pg/ml | 4.8 (1.3) | 4.1 (1.0)

4. Secondary Outcome: Interleukin-8
Description: Interleukin-8 an inflammatory cytokine which will be releases after LPS treatment.
Time Frame: measured in LPS treated blood before and after 3 weeks of Rosuvastatin treatment
Population: 16 subjects that met the inclusion/exclusion criteria the pre-post analysis allowed the use of paired T-test
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Pre-Treatment IL-8: IL-8 concentrations in blood treated with LPS before treatment with rosuvastatin
- Post-treatment IL-8: IL-8 concentrations in blood treated with LPS after treatment with rosuvastatin
Arm/Group | Pre-Treatment IL-8 | Post-treatment IL-8
Number analyzed (Participants) | 16 | 16
pg/ml | 155 (45) | 125 (27)

ADVERSE EVENTS:
Time Frame: Collected over 3 weeks for each subject
Groups:
- Rosuvastatin: Single arm non-therapeutic study
Arm/Group | Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=16)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
insomnia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes